CLINICAL TRIAL: NCT00790777
Title: A Single-dose, Open-label, Randomized, 2-way Crossover Pivotal Bioequivalence Study of 12 mg Paliperidone Extended Release Tablets Manufactured at Gurabo and Vacaville Under Fasted Condition in Healthy Subjects
Brief Title: A Study of the Bioequivalence of 12 mg Paliperidone Extended Release Tablets Manufactured at Gurabo and Vacaville
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR012085
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia
Keywords: Paliperidone ER; Schizophrenia, Mood disorders, Antipsychotic drugs
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to establish bioequivalence of paliperidone ER tablets manufactured at Gurabo as compared to paliperidone ER tablets manufactured at Vacaville, administered as a single dose of 12 mg under fasted conditions to healthy male volunteers, and to assess the safety and tolerability of both formulations.

DETAILED DESCRIPTION:
This is a randomized, open-label, 2-way crossover study in healthy male adults.The study consists of a screening phase and an open label treatment phase during which each patient will receive the 2 treatments of the study drug separated by a washout period of 7 to 14 days. Treatment A will consist of a single oral dose of 12-mg paliperidone ER, tablets manufactured at Gurabo, administered under fasted condition. Treatment B will consist of a single oral dose of 12-mg paliperidone ER, tablets manufactured at Vacaville, administered under fasted condition. Blood samples for pharmacokinetic analysis will be collected at pre-dose and for 96 hours post-dose for each period. As a change in manufacturing site will take place, bioequivalence between 12 mg tablets (highest dose strength) from the 2 production sites (Gurabo [Puerto Rico, USA] and Vacaville [California, USA]) needs to be demonstrated. This pivotal bioequivalence study is designed to examine the pharmacokinetics, safety, and tolerability of paliperidone ER manufactured at Gurabo in comparison with paliperidone ER manufactured at Vacaville

Two single oral doses of paliperidone ER 12 mg

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (weight [kg]/height [m2]) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the patient is supine for 5 minutes) between 100 and 140 mmHg systolic, inclusive, and between 50 and 90 mmHg diastolic
* Non-smoker

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the volunteer
* History of any cancer, with the exception of basal cell carcinoma
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening or at admission to the study center
* At screening, has signs of autonomic dysfunction as indicated by a decrease of > 20 mmHg in systolic blood pressure or a decrease of > 10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <40 bpm) as determined by screening 12-lead ECG
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen) or ibuprofen, within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a volunteer has a history of, drug or alcohol abuse and/or dependence within the past 5 years
* Known history of drug-induced dystonia or Neuroleptic Malignant Syndrome
* Positive test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies
* History of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or volunteer's verbal report

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To establish bioequivalence of paliperidone ER tablets manufactured at Gurabo compared with paliperidone ER tablets manufactured at Vacaville, administered as a single oral dose of 12 mg under fasted conditions

SECONDARY OUTCOMES:
To asses the safety and tolerability of both formulations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the bioequivalence of 12 mg paliperidone extended release tablets manufactured at Gurabo and Vacaville — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=741&filename=CR012085_CSR.pdf